CLINICAL TRIAL: NCT05859542
Title: Place of the Video-laryngoscope in Learning Intubation by Simulation
Status: Completed | Type: Observational
Sponsor: Mongi Slim Hospital (Other)
Responsible Party: Principal Investigator, Mhamed Sami Mebazaa, Professor, Mongi Slim Hospital
Other Study IDs: Sim intubation
Record Dates: First submitted 2023-04-30; First posted 2023-05-16 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Airway Management; Intubation, Intratracheal; Simulation; Laryngoscopy

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: The group A included 18 trainees, who started the session with videolaryngoscope followed by the direct laryngoscope.
  Interventions: Device: Videolaryngoscope first
- Group B: The group B included 17 trainees, who started the session with the direct laryngoscope followed by the videolaryngoscope.
  Interventions: Device: Direct laryngoscope first

INTERVENTIONS:
Device: Videolaryngoscope first — started the session with 3 intubations using the videolaryngoscope
  Other Names: VL
  Groups: Group A
Device: Direct laryngoscope first — started the session with 3 intubations using the Direct laryngoscope
  Other Names: DL
  Groups: Group B

SUMMARY:
The aim of the study was to determine the impact of the videolaryngoscope on reducing the time needed to intubate on a low-fidelity manikin for beginners.

The investigators conducted a randomised crossover study, which took place in the simulation department of the medical school of Tunis. They used a low-fidelity manikin designed for learning airway management. The first part of our session consisted in a theoretical training. The second part was the practical training with procedural simulation.

DETAILED DESCRIPTION:
Simulation is nowadays a widespread teaching method, particularly in airway management. The direct laryngoscope is the most commonly used device for learning intubation. As for the videolaryngoscope, it is mostly used on an advanced level, for teaching difficult laryngoscopy to professionals. Its impact on teaching intubation to beginners remains unclear.

The aim of the study was to determine the impact of the videolaryngoscope on reducing the time needed to intubate on a low-fidelity manikin for beginners.

The investigators conducted a randomised crossover study, which took place in the simulation department of the medical school of Tunis. They used a low-fidelity manikin designed for learning airway management. They included 35 trainees.

The first part of our session consisted in a theoretical training, during which one single instructor exposed the anatomical basis and the material needed: a direct laryngoscope (Macintosh) with a number 3 curved blade, a videolaryngoscope (Med-Captain) with a number 3 curved blade and a number 7 tracheal tube with a stylet.

The second part was the practical training with procedural simulation. The investigators randomized the trainees in two groups.

Each trainee proceeded to three intubations with each device, in the specified order.

The investigators used the SPSS software for data analysis. The investigators considered a p-value < 0.05 as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* fifth year's medical students.
* consentment of the participants

Exclusion Criteria:

* participants who had previously performed a tracheal intubation.

Ages: 22 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: We included 35 trainees. they were aged between 22 and 24 years old.
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-06-27 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
the time needed for the first intubation. | up to 2 minutes
  Time en seconds needed for the tube to pass through the vocal cords.

SECONDARY OUTCOMES:
the Cormack-Lehane grade | up to 2 minutes
  Cormack and Lehane grades (1 to 4)
the satisfaction of the trainees. | up to 24 hours
  The score of satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Mhamed Sami MS Mebazaa, Pr, Principal Investigator — Mongi Slim Hospital
Locations (1):
- Mongi Slim hospital, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided